CLINICAL TRIAL: NCT04653324
Title: The FARE Patient Registry: A Registry for the Food Allergy Community
Brief Title: A Registry for the Food Allergy Community
Acronym: FPR
Status: Recruiting | Type: Observational
Sponsor: Food Allergy Research & Education (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00022715
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Food Hypersensitivity; Anaphylaxis; Eosinophilic Esophagitis; Food Sensitivity; Food Intolerance; Food Allergy in Infants
Keywords: food allergy
MeSH Terms: conditions — Food Hypersensitivity; Anaphylaxis; Eosinophilic Esophagitis; Food Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The FARE Patient Registry will serve as a prospective, observational food allergy reporting system that stores detailed health and other basic information about patients' real-world experiences with food allergies, to encourage open sharing of de-identified data and participation in clinical trials. The FARE Patient Registry intends to make and support scientific discoveries by enabling the food allergy community to participate directly in research.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with diagnosed food allergy

Exclusion Criteria:

* Individuals without food allergy

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population includes males and females of all ages with one or more food allergy or those who are at risk of food-induced anaphylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 23000 (Estimated)
Dates: Start 2017-08-24 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Create a registry to characterize the extent of food allergy, its etiology and other factors that contribute to disease development. | 2023

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bufford, MS, Principal Investigator — Food Allergy Research & Education
Locations (1):
- Food Allergy Research & Education, McLean, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fierstein JL, Brown D, Gupta R, Bilaver L. Understanding Food-Related Allergic Reactions Through a US National Patient Registry. J Allergy Clin Immunol Pract. 2021 Jan;9(1):206-215.e1. doi: 10.1016/j.jaip.2020.08.011. Epub 2020 Aug 22. PMID 32841746
- [Background] Oriel RC, Waqar O, Sharma HP, Casale TB, Wang J. Characteristics of Food Allergic Reactions in United States Restaurants. J Allergy Clin Immunol Pract. 2021 Apr;9(4):1675-1682. doi: 10.1016/j.jaip.2020.12.018. Epub 2020 Dec 15. PMID 33338685
- [Background] Gupta RS, Sehgal S, Brown DA, Das R, Fierstein JL, Casale TB, Nowak-Wegrzyn AH, Bilaver LA. Characterizing Biphasic Food-Related Allergic Reactions Through a US Food Allergy Patient Registry. J Allergy Clin Immunol Pract. 2021 Oct;9(10):3717-3727. doi: 10.1016/j.jaip.2021.05.009. Epub 2021 May 24. PMID 34033980
- [Derived] Casale TB, Warren C, Gupta S, Schuldt R, Wang R, Iqbal A, Seetasith A, Gupta R. The mental health burden of food allergies: Insights from patients and their caregivers from the Food Allergy Research & Education (FARE) Patient Registry. World Allergy Organ J. 2024 Mar 23;17(4):100891. doi: 10.1016/j.waojou.2024.100891. eCollection 2024 Apr. PMID 38559493
- [Derived] Warren C, Gupta R, Seetasith A, Schuldt R, Wang R, Iqbal A, Gupta S, Casale TB. The clinical burden of food allergies: Insights from the Food Allergy Research & Education (FARE) Patient Registry. World Allergy Organ J. 2024 Mar 15;17(3):100889. doi: 10.1016/j.waojou.2024.100889. eCollection 2024 Mar. PMID 38523669